CLINICAL TRIAL: NCT04927624
Title: Comparison of Postoperative Analgesic Efficiency of Transversus Abdominis Plane Block and Quoadratus Lumborum Block on Infants Who Underwent Single Sided Inguinal Hernia Repair: A Randomised Controlled Trial
Brief Title: Transversus Abdominis Plane Block Versus Quoadratus Lumborum Block on Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pinar Ay Sayin, specialist medical doctor, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 33334
Record Dates: First submitted 2021-06-09; First posted 2021-06-16 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Transversus Abdominis Plane Block; Quoadratus Lumborum Block
Keywords: infant; analgesic efficiency; Regional anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transversus abdominis plane (Active Comparator): In the group in which Transversus Abdominis Plan Block was applied, the patient was placed in the supine position. After skin antisepsis was achieved with 10% povidone iodine, the USG probe was placed transversely between the iliac crest and the anterolateral abdominal wall. After visualizing the external-internal obliq and transversus abdominis muscles, 0.5 ml/kg of 0.25% bupivacaine was injected after negative aspiration by advancing the needle into the fascia between the internal obliq muscle and the transversus abdominis muscle with the in-plane technique.
  Interventions: Procedure: transversus abdominis plane block
- quoadratus lumborum block (Active Comparator): In the Quadratus Lumborum Block (Lateral approach) group, the patient was placed in the lateral position with the side to be blocked on top. After skin antisepsis was achieved with 10% povidone iodine, the USG probe was placed transversely between the iliac crest and costa edge. After visualizing the extarnal-internal obliq and transversus abdominis muscles, the probe was advanced posteriorly. Quadratus lumborum muscle and thoracolumbar fascia were visualized. The needle was advanced to the anterolateral border of the quadratus lumborum muscle with the in-plane technique and 0.5 ml/kg of 0.25% bupivacaine was injected after negative aspiration.
  Interventions: Procedure: quoadratus lumborum block

INTERVENTIONS:
Procedure: transversus abdominis plane block — The transversus abdominis plane (TAP) block was first introduced by Rafi et al. in 2001 as a landmark-guided technique via the triangle of Petit to achieve a field block. It involves the injection of a local anesthetic solution into a plane between the internal oblique muscle and transversus abdominis muscle. Since the thoracolumbar nerves originating from the T6 to L1 spinal roots run into this plane and supply sensory nerves to the anterolateral abdominal wall , the local anesthetic spread in this plane can block the neural afferents and provide analgesia to the anterolateral abdominal wall.
  Other Names: quoadratus lumborum block
  Arms: transversus abdominis plane
Procedure: quoadratus lumborum block — quoadratus lumborum block
  Arms: quoadratus lumborum block

SUMMARY:
we aimed to compare the effects of TAPB and QLB on postoperative pain score and analgesic consumption in infants who underwent unilateral inguinal hernia surgery.

DETAILED DESCRIPTION:
Infants are more sensitive to the side effects of general anesthesia than older children. This may be associated with the incomplete maturation of organ systems effective in pharmacodynamics. Regional anesthesia applications provide safe and effective analgesia by reducing the need for opioids. Regional anesthesia applications in infants require experience and complication rates due to central blocks are high. However, in recent years, the use of ultrasound (USG) has increased the use of safe and effective trunk blocks. There are studies on the use of Transversus Abdominis Plan Block (TAPB) and Quadratus Lumborum Block (QLB) in children. However, there is no comparative study on its use in infants.

In our study, we aimed to compare the effects of TAPB and QLB on postoperative pain score and analgesic consumption in infants who underwent unilateral inguinal hernia surgery.

ELIGIBILITY:
Inclusion Criteria:

* 1 month to 1 year
* who were scheduled for unilateral inguinal hernia operation
* American Society of Anesthesiologists (ASA) physical score I-II

Exclusion Criteria:

* Patients with ASA II-IV
* coagulopathy
* skin infection at the block application site
* bupivacaine allergy
* bilateral inguinal hernia operation
* additional operation in different region
* laparoscopic inguinal hernia operation
* younger than 1 month
* with a history of prematurity

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — infants
Enrollment: 60 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-10-15 (Estimated)

PRIMARY OUTCOMES:
FLACC | up to 24 hours
  Face, Legs, Activitiy, Cry, Consolability score
first analgesic need times | up to 24 hours
  time of first analgesic need after surgery

SECONDARY OUTCOMES:
frequency of need for analgesics | up to 24 hours
  Frequency of analgesic requirement in the first 24 hours after the operation
complications | up to 24 hours
  post-operative anesthetic complications

CONTACTS AND LOCATIONS:
Locations (1):
- Sisli Etfal Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No